CLINICAL TRIAL: NCT02603016
Title: Phase 1 Study of Clinical Nutrition That Research Safty and Efficacy in Lung Neoplasms And Breast Carcinoma
Brief Title: Efficacy Study of Clinical Nutrition to Treat Lung Neoplasms And Breast Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhiyong Wu, Associate Chief Physician, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PLAGHS201503601
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Lung Neoplasms; Breast Neoplasms
Keywords: Clinical Nutrition
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GLSE compound group (Experimental): GLSE compound 2g each time by mouth,twice a day for 42 days.
  Interventions: Drug: GLSE compound
- Maitake mushroom extract compound group (Experimental): Maitake mushroom extract compound 2 tables each time by mouth,twice a day for 42 days.
  Interventions: Drug: Maitake mushroom extract compound
- Ginseng compound group (Experimental): Ginseng compound 2 tables each time by mouth,twice a day for 42 days.
  Interventions: Drug: Ginseng compound
- blank control group (No Intervention): Take nothing.

INTERVENTIONS:
Drug: GLSE compound
  Arms: GLSE compound group
Drug: Maitake mushroom extract compound
  Arms: Maitake mushroom extract compound group
Drug: Ginseng compound
  Arms: Ginseng compound group

SUMMARY:
This study evaluates the efficacy of clinical nutrition to treat lung neoplasms and breast carcinoma.We estimate there will be 480 patients accepted.120 patients will receive GLSE compound,120 patients will recrive Maitake mushroom extract compound,120 patients will recrive Rinseng compound,and 120 patients will be as blank countrol group.Efficacy Study of Clinical Nutrition to Treat Lung Neoplasms And Breast Carcinoma

DETAILED DESCRIPTION:
GLSE compound、Maitake mushroom extract compound and Rinseng compound have different mechanism on enhancing immunity.This clinicaltrial compare them the immune effect in the progress of treating lung neoplasms and breast carcinoma.Within the 42 days,we will abide by the plan to evaluate the immunity enhancement by monitoring mmune effector molecules.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer and breast cancer patients confirmed by surgery pathology;
* ECOG physical stamina score of 0~3 points;
* Expected lifetime > 3 months;
* Need to receive radiation and chemotherapy;
* Heart, liver and kidney function and blood picture is normal,WBC≥4×109/L, neutrophil count≥ 2 x 109 / L,platelet count≥100×109/L, hemoglobin≥100 g/L;
* To follow-up, good adherence

Exclusion Criteria:

* Allergic to text drug;
* Pregnancy or lactation women;
* Suffering from mental illness of not easy to control,
* Have serious mental or cognitive dysfunction;
* Can not comply with the experimental scheme or can't cooperate with the follow-up;
* The patients who are unfavorable to the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
T-lymphocyte cell subsets | three mouths
  T-lymphocyte cell subsets contains CD3+、CD4+、CD8+、CD28-、CD28+、CD4+CD25+、HLADR+、HLADR-,measured these cells concentration level

CONTACTS AND LOCATIONS:
Overall Officials: Shunchang Jiao, Doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- PLA general hospital, Beijing, Beijing Municipality, China